CLINICAL TRIAL: NCT00455637
Title: A Phase II, Randomised, Double-blind, Dose-ranging Study in Children and Young People to Determine the Optimal Dose of Botulinum Toxin Type-A (Dysport®) in Managing the Symptoms of Hip Muscle Spasticity Due to Cerebral Palsy
Brief Title: Which is the Best Dose of Dysport in Helping With Hip Pain for Children With Cerebral Palsy?
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low levels of recruitment
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Y-97-52120-727; 2005-001794-10 (EudraCT Number)
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dysport 5 units (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Dysport 10 units (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Dysport 15 units (Experimental)
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of the study is to compare the effectiveness of 3 doses of Dysport (5, 10 or 15 Units/Kg/hip) in the management of chronic bilateral hip pain due to cerebral palsy in children/young people.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 4 and 16 years (inclusive).
* Diagnosis of cerebral palsy.
* Presence of clinical bilateral hip pain (of at least 6 months duration) due to cerebral palsy as defined by the child/young person and/or parents.
* Paediatric Pain Profile score of 25 or greater.

Exclusion Criteria:

* Prior treatment with Botulinum toxin (any serotype, administered anywhere in the body) within 4 months prior to Screening.
* Planned or anticipated requirement for surgery during the study period.
* History of hypersensitivity to the investigational drug or any of its excipients.
* Likely to require treatment during the study with drugs that are not permitted by the study protocol or that in the opinion of the Investigator may interfere with the evaluation of the efficacy or safety of the study medication.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03-17 (Actual); Study Completion 2008-03-17 (Actual)

PRIMARY OUTCOMES:
To compare the effectiveness of 3 doses of Dysport (5, 10 or 15 Units/Kg/hip) in the management of chronic bilateral hip pain due to cerebral palsy in children/young people. | From baseline to the end of study (week 20)
The primary endpoint will be the change in score in the Paediatric Pain Profile. | From baseline to the week 4 assessment

SECONDARY OUTCOMES:
To compare the effectiveness of 3 doses of Dysport (5, 10 or 15 Units/Kg/hip) in the management of hip pain as assessed by the change in the score of the Paediatric Pain Profile at all other assessment time points. | Weeks 12, 16 and 20
To compare the effect of the different doses of Dysport on sleep pattern and quality as assessed using a sleep diary and sleep questionnaire at all assessment time points. | Weeks 4, 12, 16 and 20
To compare the effect of the different doses of Dysport on oral analgesia intake for hip pain at all assessment time points. | Weeks 4, 12, 16 and 20

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Chailey Heritage Clinical Services, Chailey, United Kingdom